CLINICAL TRIAL: NCT07222384
Title: A PHASE 3 PROTOCOL TO INVESTIGATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A BNT162b2 (LP.8.1)-ADAPTED VACCINE IN CHILDREN 5 THROUGH 11 YEARS OF AGE CONSIDERED AT HIGH RISK FOR SEVERE COVID-19
Brief Title: A Study to Learn About BNT162b2 (LP.8.1)-Adapted Vaccine Against SARS-CoV-2 in Children 5 Through 11 Years of Age That Are Considered at Higher Risk of Severe COVID-19
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: C4591082
Record Dates: First submitted 2025-10-28; First posted 2025-10-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: COVID-19; SARS-COV-2 Infection
Keywords: Respiratory Tract Infections; Infections; Virus Diseases; Coronavirus Infections; Coronaviridae Infections; Lung Diseases; Respiratory Tract Diseases; COVID-19; mRNA Vaccines; Nucleic Acid-Based Vaccines; Vaccines; Biological Products; COVID-19 Vaccines; Viral Vaccines; Antigens; Biological Factors; BNT162 Vaccine
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections; Infections; Virus Diseases; Coronavirus Infections; Coronaviridae Infections; Lung Diseases; Respiratory Tract Diseases | interventions — BNT162 Vaccine

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 5-11 Years (Higher-Risk Individuals) (Experimental): BNT162b2 (2025/2026 formulation)
  Interventions: Biological: BNT162b2 (2025/2026 formulation)

INTERVENTIONS:
Biological: BNT162b2 (2025/2026 formulation) — BNT162b2 (formulation targeting the 2025/2026 recommended SARS-CoV-2 strain)

SUMMARY:
The purpose of this study is to learn about the safety, tolerability, and immunogenicity of an updated vaccine against COVID-19, called BNT162b2 (2025/2026 formulation).

This study is seeking participants 5 through 11 years of age who:

* have at least 1 underlying condition that puts them at high risk for severe outcomes from COVID-19,
* and are medically stable.

All participants in this study will receive 1 vaccine dose given in the muscle of their arm of a BNT162b2 (2025/2026 formulation) vaccine which targets the COVID-19 virus, specifically the strain selected for the 2025-2026 COVID-19 viral respiratory season.

Participants will take part in this study for about 6 months and will need to visit the clinical study site at least 2 times.

ELIGIBILITY:
Key Inclusion Criteria:

* Children 5 through 11 years of age at their first appointment.
* Children with at least 1 underlying stable medical condition that increases their risk of severe COVID-19, as listed in the protocol.

Key Exclusion Criteria:

* Children who have had confirmed COVID-19 within the last 5 months (150 days).
* Children who have received a COVID-19 vaccine, either as part of a research study or an approved vaccine, within the last 5 months (150 days).
* Children who have received a 2025-2026 seasonal COVID-19 vaccination.
* Children with a history of myocarditis or pericarditis.
* Children with a previous or current diagnosis of Multisystem Inflammatory Syndrome in Children (MIS-C)
* Children with a medical condition wherein they would be considered for a second dose of COVID-19 vaccine to protect against risk of severe COVID-19 based on standard of care.

Refer to the study contact for further eligibility details.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 343 (Actual)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting local reactions | For up to 7 days after vaccination
Percentage of participants reporting systemic events | For up to 7 days after vaccination
Percentage of participants reporting adverse events | Through 1 month after vaccination
Percentage of participants reporting serious adverse events | Through 6 months after vaccination
Geometric Mean Fold Rises (GMFRs) | From before vaccination to 1 month after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (27):
  - Stanford University Medical Center CTRU - 800 Welch Road, Palo Alto, California
  - California Research Foundation, San Diego, California
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - C & R Research USA, Homestead, Florida
  - Florida Pharmaceutical Research and Associates, Miami, Florida
  - Bio-Medical Research LLC, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - GCP Research, Global Clinical professionals, St. Petersburg, Florida
  - Medical Research Partners, Ammon, Idaho
  - AMR Clinical, Oak Brook, Illinois
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - Michigan Center of Medical Research (MICHMER), Bingham Farms, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - University of Rochester Medical Center, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - DM Clinical Research- Cyfair, Houston, Texas
  - ACRC Trials, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Javara - Privia Medical Group North Texas - Stephenville, Stephenville, Texas
  - AMR Clinical, Layton, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Tekton Research, LLC., Richmond, Virginia
- Puerto Rico (2):
  - Clinical Research Puerto Rico, Guayama
  - Ponce Medical School Foundation Inc., Ponce

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591082